CLINICAL TRIAL: NCT00720317
Title: Diabetic Retinopathy and Sickle Cell Trait
Brief Title: Diabetic Retinopathy and Sickle Trait
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Esther M. Bowie, MD, Medical University of South Carolina
Other Study IDs: SEI-08-001
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Diabetic Retinopathy; Sickle Cell Trait
Keywords: Diabetic Retinopathy; Sickle Cell Trait; Vision Loss; Eye disease
MeSH Terms: conditions — Diabetic Retinopathy; Sickle Cell Trait; Vision Disorders; Eye Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To more clearly ascertain the relationship between ocular manifestations of sickle cell disease and diabetes, specifically; whether the presence of sickle cell trait exacerbates the disease progression of diabetic retinopathy.

DETAILED DESCRIPTION:
The objective of this research study is to evaluate the relationship between sickle cell trait and the progression of diabetic retinopathy. People with diabetes have high blood sugar that damages small blood vessels. Damage to the blood vessels that supply the retina in the back of the eye is called diabetic retinopathy. Diabetic retinopathy is worse in African-Americans with diabetes, with earlier and more severe disease progression and common complications including vitreous hemorrhage - where these blood vessels in the eye leak - and retinal detachment - the separation of the nerves of the retina from the back of the eye which may lead to blindness. One explanation for this increased severity of diabetes in African-Americans is the presence of sickle cell disease, or even just sickle trait, which causes damage to red blood cells and blood vessels under conditions of stress; like low oxygen levels, or hyperglycemic acidosis.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified African-American patients with diabetes will be identified from Dr Bowie's retina clinic at Storm Eye Institute.
* These subjects are either being screened or treated for the progression of diabetic retinopathy.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: African-Americans with type II diabetes mellitus experience increased systemic vascular morbidity and mortality, even after adjustment for socioeconomic factors.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
We aim to screen African-American diabetic patients with retinopathy to ascertain whether sickle trait is present, and if so whether there is increased severity of diabetic retinopathy in the group with sickle trait. | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Esther M. Bowie, MD, Principal Investigator — Medical University of South Carolina, Storm Eye Institute
Locations (1):
- Medical University of South Carolina, Storm Eye Institute, Charleston, South Carolina, United States